CLINICAL TRIAL: NCT07257133
Title: Opioid Avoidance In Surgery Through Integrating Suzetrigine: Post-Operative Care Phase Pilot
Brief Title: A Study Of Opioid Avoidance In Surgery Through Integrating Suzetrigine
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Deanna C. Menapace, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 25-004867
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Post Operative Pain
Keywords: Facial plastic surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Suzetrigine (Experimental): Patients will receive Suzetrigine in place of opioid medications for post-operative pain management.
  Interventions: Drug: Suzetrigine

INTERVENTIONS:
Drug: Suzetrigine — Patients will receive suzetrigine instead of the standard of care opioids.
  The dosing schedule will be: a single oral loading dose of 100 mg suzetrigine, followed by 50 mg every 12 hours starting 12 hours after the first dose. Treatment will begin right after surgery and continue for up to 7 days.
  All patients will also receive acetaminophen (650 mg every 6 hours) and celecoxib (200 mg every 24 hours) as part of the standard multimodal pain management regimen.
  Patients experiencing breakthrough pain will be prescribed rescue opioid medication (oxycodone 5 mg every 6 hours as needed) and use will be recorded.

SUMMARY:
This prospective, single-arm feasibility study will evaluate postoperative pain control, opioid use, and early recovery outcomes in adult patients undergoing elective outpatient facial plastic surgery who receive suzetrigine as part of their standard postoperative analgesic regimen.

DETAILED DESCRIPTION:
Traditional postoperative pain management in facial plastic surgery often relies on opioid analgesics. While effective, their use is associated with adverse effects such as constipation, nausea, vomiting, sedation, respiratory depression, and dependency risk. In the context of the ongoing opioid misuse public health crisis, identifying effective non-opioid alternatives is crucial.

Suzetrigine is a first-in-class oral analgesic that selectively inhibits the voltage-gated sodium channel NaV1.8. These channels are selectively expressed within peripheral pain-sensing neurons and do not have a functional role within the central nervous system (CNS). Unlike opioids, suzetrigine does not cross the blood-brain barrier and avoids CNS side effects such as sedation, respiratory depression, and addiction potential.

In January 2025, the U.S. Food and Drug Administration (FDA) approved suzetrigine for the short-term treatment of moderate-to-severe acute pain in adults. Approval was supported by two Phase 3 randomized controlled trials in patients undergoing abdominoplasty (NCT05558410) and bunionectomy (NCT05553366), both standard models for acute postoperative pain. In these studies, suzetrigine demonstrated analgesic efficacy comparable to hydrocodone/acetaminophen, with a faster onset of meaningful pain relief than placebo and a favorable tolerability profile.

Despite this evidence, there is currently no data on the use of suzetrigine in facial plastic surgery. The integration of suzetrigine into postoperative pain management regimens for this population has the potential to reduce opioid prescription patterns and improve patient outcomes. This single-arm feasibility study aims to describe our early experience with suzetrigine and provide preliminary evidence to inform the feasibility and design of future prospective trials.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) undergoing elective outpatient facial plastic surgery.
* Able to consent and comply with study procedures.
* Planned postoperative use of suzetrigine per provider discretion.

Exclusion Criteria:

* Age <18.
* Pregnant or breastfeeding.
* Women on hormonal birth control who decline suzetrigine-related counseling.
* Patients using strong CYP3A4 inhibitor medications (i.e. itraconazole, ketoconazole, clarithromycin, ritonavir, and grapefruit juice).
* Known allergy to suzetrigine.
* Vulnerable or protected research populations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Total opioid consumption | 7 days post-operation
  Number of opioid pills used during the first 7 postoperative days
Number of patients with no rescue use | 7 days post-operation
  Total number of patients who do not use any rescue opioids postoperatively

SECONDARY OUTCOMES:
Pain intensity score | 1 day post-operation
  Pain intensity score during the first postoperative day will be measured by the 1 question Visual Analog Scale for pain. Patients will rank level of pain experienced on a 10 point Likert scale, with 0 = No pain and 10 = Worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Deanna C. Menapace, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No